CLINICAL TRIAL: NCT01173822
Title: Processed Residual Pump Blood in Cardiac Surgery: The PRBC Trial
Acronym: PRBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Dr. Richard Whitlock, Population Health Research Institute
Organization: McMaster University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PRBC-1
Record Dates: First submitted 2010-07-16; First posted 2010-08-02 (Estimated); Last update posted 2010-08-02 (Estimated); Status verified 2010-07

CONDITIONS: Cardiopulmonary Bypass; Hemorrhage; Surgery
Keywords: cardiopulmonary bypass; hemorrhage; trials; surgery
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): Ultra filtration of residual blood.
  Interventions: Other: Ultrafiltration of residual blood
- Control (No Intervention): The current practice in our institution was to displace all the remaining volume in the CPB circuit into a transfer pack by displacing the remaining blood in the CPB circuit with additional Lactated Ringers solution. This transfer pack is then given to the anesthetist for reinfusion into the patient.
  Interventions: Other: Ultrafiltration of residual blood

INTERVENTIONS:
Other: Ultrafiltration of residual blood — The inflow line to the hemoconcentrator was connected to the sideport of the arterial filter stopcock, allowing the residual blood in the CPB circuit to be processed through the hemoconcentrator. The outflow line from the hemoconcentrator was connected to a second three way stopcock located on the cardiotomy reservoir. Blood was circulated from the venous reservoir through the hemoconcentrator and returned to the venous reservoir until the desired hematocrit was achieved. The blood was then diverted to a transfer pack until all the blood from the venous reservoir, heat exchanger, and membrane oxygenator had been filtered and hemoconcentrated. This transfer pack was given to the anesthetist for reinfusion into the patient.

SUMMARY:
The study is an randomized controlled trial (RCT) of 198 coronary artery bypass graft (CABG) patients, exploring whether ultrafiltration of residual blood in the cardiopulmonary bypass circuit reduces transfusion and bleeding.

DETAILED DESCRIPTION:
Blood products are a limited resource and cardiac surgery is a high consumer. Processing residual cardiopulmonary bypass (CPB) volume via ultrafiltration may improve hemostasis and reduce transfusion through clearing activated complement, activated coagulation components, and proinflammatory cytokines. Unlike cell saver technology, ultrafiltration has the advantage of maintaining plasma proteins, platelets, and coagulation factors. We sought to establish if the processing of residual CPB volume with ultrafiltration reduces homologous blood transfusion and bleeding.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* were to undergo isolated on-pump CABG
* were able to give informed consent

Exclusion Criteria:

* performed autologous blood donation
* underwent off-pump CABG
* emergency procedure
* resternotomy
* known bleeding disorder not drug related
* history of heparin-induced thrombocytopenia
* Jehovah's Witness
* intra-operative catastrophe prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-12; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
the proportion of patients transfused with homologous red blood cells (RBC) | At 30 days post-operatively

SECONDARY OUTCOMES:
Proportion of patients transfused with any blood product | At 30 days post-operatively
Volume of pRBC's transfused post-operative | At 30 days post-operatively
Post-operative hemorrhage | At 24 hours post-operative
Discharge Hemoglobin | A date of discharge, median 5 days in study
Length of hospital stay | From day to surgery to discharge, median 5 days in this study

CONTACTS AND LOCATIONS:
Overall Officials: Richard Whitlock, MD MSc, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Whitlock R, Mathew J, Eikelboom J, Al-Saleh AM, Yuan F, Teoh K. Processed residual pump blood in cardiac surgery: the Processed Residual Blood in Cardiac surgery trial. Transfusion. 2013 Jul;53(7):1487-92. doi: 10.1111/j.1537-2995.2012.03958.x. Epub 2012 Nov 26. PMID 23176311